CLINICAL TRIAL: NCT01233739
Title: Chondroitin Sulphate Treatment Efficacy in Rhizarthrosis. Measurement With Sensory and Quantitive Functional Tests and Concordance Analysis With Subjective Scales of Pain.
Brief Title: Chondroitin Sulphate Treatment Efficacy in Rhizarthrosis.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Juan A. Arnaiz (Other)
Responsible Party: Sponsor-Investigator, Juan A. Arnaiz, MD, PhD, Hospital Clinic of Barcelona
Organization: Hospital Clinic of Barcelona (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RIZACONDRO
Record Dates: First submitted 2010-11-02; First posted 2010-11-03 (Estimated); Last update posted 2013-02-22 (Estimated); Status verified 2013-02

CONDITIONS: Rhizarthrosis
Keywords: rhizarthrosis; Chondroitin sulfate; Placebo
MeSH Terms: interventions — Chondroitin Sulfates

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Chondroitin sulfate (Experimental): Administration of 2 capsules of 400 mg of chondroitin sulfate orally.
  Interventions: Drug: Chondroitin sulfate

INTERVENTIONS:
Drug: Chondroitin sulfate — Administration of 2 capsules of 400 mg of chondroitin sulfate orally.
  Arms: Chondroitin sulfate
Drug: Placebo — Administration of 2 capsules of placebo orally.
  Arms: Placebo

SUMMARY:
Patients who present rhizarthrosis diagnostic will be randomized to be treated with chondroitin sulfate or placebo during 24 weeks to study the effect of the treatment with objective and subjective indicators of pain and sensibility.

ELIGIBILITY:
Inclusion Criteria:

* both sex patients
* age between 45 to 75 years
* with mechanical pain at the trapezium-thumb metacarpal joint of more than 3 months duration
* grade II or III Eaton & Glickel rhizarthrosis radiological diagnose
* pain at inclusion of >= 40 mm at a visual analogue scale
* without rehabilitation treatment or infiltration in the last 6 months
* who accept to participate and sign informed consent

Exclusion Criteria:

* patients with rhizarthrosis resulted from rheumatic disease
* patients with joint surgery or traumatic background
* illiterate patients or unable to understand informed consent
* patients with previous neuropsychopathology enough severe to unable participation at the study
* patients with peripheral sensory impairment due to diabetes, peripheral neuropathy or central neurological sequelae of disease in the affected limb that can alter sensory perception
* patients with coagulopathy
* inflammation for other process at the joint at study
* in treatment with non-steroidal anti-inflammatory drug in the last 7 days and/or corticosteroid in the last 30 days
* allergy or hypersensibility at chondroitin sulfate or its excipients
* pregnant or breastfeeding woman

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2011-03; Primary Completion 2013-04 (Estimated); Study Completion 2013-04 (Estimated)

PRIMARY OUTCOMES:
Evaluation with visual analogue pain scale as mean at the last weak | 36 weeks

SECONDARY OUTCOMES:
Sollerman test | 36 weeks
  Evaluation of hand function with Sollerman test
Hand pressure force | 36 weeks
Thumb-index finger pincer force | 36 weeks
Dash test | 36 weeks
  Osteoarthritis functional test
SF-12 test | 36 weeks
  Quality of life test
Mechanical sensitivity measured with electronic Von Frey filament | 36 weeks
vibratory and thermic sensibility threshold assisted by computer | 36 weeks
Use of paracetamol or other analgesic drugs | 36 weeks
  recorded in a patient diary
Evolution of trapezium-thumb metacarpal joint by ultrasound scan | 36 weeks
Hematologic evaluation | 24 weeks
Biochemical evaluation | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Joaquím Forés, MD, Principal Investigator — Hospital Clínic i Provincial de Barcelona
Locations (1):
- Hospital Clínic i Provincial de Barcelona, Barcelona, Catalonia, Spain